CLINICAL TRIAL: NCT03288012
Title: Sickle Cell Disease: Targeting Alloantibody Formation Reduction; Risk Factors, and Genetics
Acronym: STARRING
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sanquin Research & Blood Bank Divisions (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Radboud University Medical Center (Other); HagaZiekenhuis (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL60834.018.17
Record Dates: First submitted 2017-09-13; First posted 2017-09-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2018-08

CONDITIONS: Alloimmunization; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for DNA analysis and analysis of immune system components involved in alloimmune reactions following erythrocyte transfusion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The focus of the study is the pathophysiological mechanism of allo-antibody formation after red blood cell transfusion in sickle cell disease patients.

DETAILED DESCRIPTION:
The main objectives of this study are to study the role of the innate and adaptive immune response in allo-antibody formation and furthermore to identify the genetic and time dependent clinical risk factors on alloimmunization in SCD patients.

Subjects without allo-antibodies, receiving a red blood cell transfusion, will be included in this study. At 5 time points blood will be drawn from these subjects. (T0: Before transfusion, T1: 1 day after transfusion, T2: 1 week after transfusion, T3: 4 weeks after transfusion, T4: 6 months after transfusion).

At each time point specific markers of the immune system will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease
* Receiving a red blood cell transfusion

Exclusion Criteria:

* Previous positive screen for allo-antibodies
* >25 red blood cell units in the past

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sickle cell disease population receiving care in the participating hospitals
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The innate and adaptive immune response of patients with sickle cell disease that form allo-antibodies following erythrocyte transfusion, compared to patients that do not form alloantibodies following erythrocyte transfusion | 6 months
  Multiple activating and regulatory markers of the innate and adaptive immune system will be measured at the indicated time points and compared between cases and controls

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Academic Medical Center Amsterdam, Amsterdam-Zuidoost
  - Radboudumc, Nijmegen
  - Erasmus MC, Rotterdam
  - HagaZiekenhuis, The Hague